CLINICAL TRIAL: NCT05813912
Title: Protocol Title: A Single Arm Study Investigating the Glycaemic Control and Safety of Adding Semaglutide to Insulin Icodec in Participants With Type 2 Diabetes Qualifying for Treatment Intensification Short Title: A Research Study to See How a New Weekly Insulin, Insulin Icodec When Given Along With Semaglutide Helps in Reducing the Blood Sugar Level in Patients With Type 2 Diabetes
Brief Title: A Research Study to See How a New Weekly Insulin, Insulin Icodec When Given Along With Semaglutide Helps in Reducing the Blood Sugar Level in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4910; 2022-002847-24 (EudraCT Number); U1111-1281-4752 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Insulin Icodec + Semaglutide (Experimental): Participants will receive insulin icodec once weekly for 26 weeks in run-in period to ensure the dose optimization. Thereafter, participants meeting intensification criteria will proceed to the 26-week treatment period to receive once weekly semaglutide subcutaneously starting from 0.25 milligrams (mg) and dose increased up to 1 mg along with 700 units per milliliter (U/mL) insulin icodec therapy. There are no maximum or minimum insulin doses.
  Interventions: Drug: Insulin Icodec; Drug: Semaglutide

INTERVENTIONS:
Drug: Insulin Icodec — Participants will receive subcutaneously insulin icodec once weekly for 52 weeks.
Drug: Semaglutide — Participants will receive once weekly semaglutide subcutaneously starting from 0.25 mg and dose increased up to 1 mg for 26 weeks.

SUMMARY:
This study looks at how a new medicine insulin icodec helps in reducing blood sugar levels when given along with semaglutide in patients with type 2 diabetes. Participants will get the medicine insulin icodec once a week in the first part of the study (run-in period-26 weeks). Participants will only enter the second part of the study if the blood sugar levels have not reduced to normal. If blood sugar levels are normal after the first 26 weeks, participants will continue in a 5-week follow up period. In the second part of the study (intensification period-26 weeks), participants will get both insulin icodec and semaglutide once weekly after which they will continue in a 5-week follow up period. Participants will have to inject the study medicines once a week on the same day of the week in a skin fold in the thigh, upper arm or stomach. The study will last for about 13 months. Participants will get a blood glucose meter to check blood sugar levels. In addition, participants will be asked to enter blood sugar levels in the study phone. In addition, Participants will be asked to enter selected few blood sugar values (three times during the study) in a paper diary that will be provided to participants. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes (T2D) greater than or equal to (>=) 180 days prior to the day of screening
* HbA1c from 7.5%-10.5% (58-91 millimoles per mole [mmol/mol]) (both inclusive)
* Treated with once daily or twice daily basal insulin (minimum of 0.25 international units per kilograms per day (IU/kg/day) or 20 IU/day) without concomitant glucagon-like peptide-1 receptor agonists (GLP-1 RA) >= 90 days prior to the day of screening with or without any of the following antidiabetic drugs/regimens with stable doses >= 90 days prior to screening: metformin, sulfonylureas, meglitinides (glinides), dipeptidyl peptidase-4 (DPP-4) inhibitors, Sodium-glucose Cotransporter-2 (SGLT2) inhibitors, thiazolidinediones, alpha-glucosidase inhibitors. Oral combination products (for the allowed individual oral anti-diabetic drugs)

Exclusion Criteria:

* Presence or history of pancreatitis (acute or chronic) within 180 days before screening
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening and between screening and initiation
* Chronic heart failure classified as being in New York Heart Association (NYHA) Class IV at screening
* Planned coronary, carotid or peripheral artery revascularization
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and initiation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 52 (visit 54)
  Measured in percentage (%) points.

SECONDARY OUTCOMES:
Change in mean 7-point self-measured plasma glucose (SMPG) profiles | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 52 (visit 54)
  Measured in millimoles per liter (mmol/L).
Change in mean post-prandial glucose increment (over all meals) | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 52 (visit 54)
  Measured in mmol/L.
Change in fasting plasma glucose (FPG) | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 52 (visit 54)
  Measured in mmol/L.
Number of severe hypoglycaemic episodes (level 3) | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 57 (visit 56)
  Measured in number of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (less than [<] 3.0 mmol/L [54 milligrams per deciliter {mg/dL}], confirmed by blood glucose [BG] meter) | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 57 (visit 56)
  Measured in number of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L [54 mg/dL]), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 57 (visit 56)
  Measured as number of episodes.
Change in body weight | From baseline (time of insulin icodec and semaglutide initiation [week 26, visit 28]) to week 52 (visit 54)
  Measured in kilograms (Kg).
Relative change in weekly insulin icodec dose | From the week prior to intensification, week 25 (visit 27) to week 52 (visit 54)
  Measured in units (U).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (29):
- Czechia (6):
  - Edumed Broumov, Broumov
  - DIALINE s.r.o., Plzeň 3
  - Diabet2 s.r.o., Prague
  - Diabetologická a endokrinologická ambulance Praha, Prague
  - EUC Klinika Praha a.s., Prague
  - Comfort Care Praha s.r.o., Praha 4 - Chodov
- Malaysia (4):
  - Hospital Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya, Putrajaya
  - Hospital Miri, Miri, Sarawak
  - Universiti Teknologi MARA, Sungai Buloh Campus, Sungai Buloh, Selangor
- Poland (12):
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Osrodek Badan Klinicznych "METABOLICA" lek. Robert Witek, Tarnów, Lesser Poland Voivodeship
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski, Lubusz Voivodeship
  - NBR Polska, Warsaw, Masovian Voivodeship
  - Osteo-Medic s.c. A. Racewicz, J. Supronik, Bialystok
  - NZOZ Gdanska Poradnia Cukrzycowa Sp.z o.o., Gdansk
  - NZOZ Gdanska Poradnia Cukrzycowa, Gdansk
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski
  - Centrum Medyczne Pratia Katowice, Katowice
  - Santa Sp. z o.o, Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - NBR Polska Tomasz Klodawski, Warsaw
  - Santa Sp. z o.o, Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz, Łódź Voivodeship
- Serbia (4):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - CHC Zvezdara, Clinical department for endocrinology, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Clinical Centre Kragujevac, Internal Diseases Clinic, Endocrinology department, Kragujevac
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com